CLINICAL TRIAL: NCT01801150
Title: Effect Of Nasal CPAP On Glycemic Control In Patients With Poorly Controlled Type 2 Diabetes And Sleep Apnea-Hypopnea Syndrome
Brief Title: CPAP in Diabetes Type 2 Patients With Sleep Apnea
Acronym: DM-SAHS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Francisco Garcia-Rio, PhD, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HULP-DM-SAHS-2012
Record Dates: First submitted 2012-11-16; First posted 2013-02-28 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Sleep Apnea
Keywords: Diabetes; Apnea- hypopnea Syndrome; Glycemic control; Prevalence; SAHS; life quality
MeSH Terms: conditions — Diabetes Mellitus; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- lifestyle and diabetes treatment (No Intervention): Counseil about lifestyle and current diabetes treatment
- CPAP nasal treatment (Experimental): Continuous positive airway pressure (CPAP) nasal during the night and current diabetes treatment. Device
  Interventions: Device: CPAP nasal treatment

INTERVENTIONS:
Device: CPAP nasal treatment — Treatment with titred CPAP nasal during the nighttime
  Arms: CPAP nasal treatment

SUMMARY:
Aim: To assess if six months of treatment with CPAP associated with conventional drug therapy, contribute to improved glycemic control in patients with type 2 diabetes and sleep apnea-hypopnea syndrome SAHS)

DETAILED DESCRIPTION:
Main objective:

To assess the effect of 6 months of CPAP treatment associated with conventional drug therapy on glycemic control in patients with type 2 diabetes and sleep apnea-hypopnea syndrome (SAHS)

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 to 75 years old; diagnosis of type 2 diabetes mellitus; treatment with diet; oral antidiabetics or insulin stable in the last month; levels of HbA1c> 7.5% (if not supported clinic two controls to confirm with a difference not exceeding 0.5%); overweight or obese (BMI ≥ 25 kg/m2)

Exclusion Criteria:

* professional drivers, risk profession or respiratory failure; excessive daytime sleepiness is very high (Epworth scale> 18); morbid obesity (BMI> 40 kg/m2); CPAP treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Six months
  To assess the effect of 6 months of CPAP therapy and conventional treatment on glycemic control in patients with type 2 diabetes and sleep apnea-hypopnea syndrome (SAHS)

SECONDARY OUTCOMES:
To determine additional effects of CPAP on insulin resistance in patients with type 2 diabetes and SAHS. | 6 months
  . Determine the medium term additional effect of CPAP on insulin resistance in patients with type 2 diabetes and SAHS.

OTHER OUTCOMES:
Impact of CPAP on glycemic control | 6 months
  Analyze the impact of additional treatment with CPAP on serum lipids and C-reactive protein concentration in patients with type 2 diabetes and SAHS
Quality of life after CPAP | 6 months
  Establish the impact of additional treatment with CPAP on quality of life related to health of patients with type 2 diabetes and SAHS.
Inflammatory markers after CPAP | 6 months
  To evaluate the effect of CPAP on inflammatory cytokines, biomarkers of oxidative stress, sympathetic tone and intake regulating hormones in patients with type 2 diabetes and SAHS.
Endocrine control with CPAP treatment | 6 months
  Relate the CPAP-induced changes in the concentration of HbA1c and HOMA index with changes produced in the basal inflammatory reaction, oxidative stress, sympathetic activity and intake regulatory hormones.
  Identify the subset of patients with poorly controlled type 2 diabetes and SAHS in the six months of treatment with CPAP achieve a more pronounced reduction in HbA1c.
Influence of body distribution and activity on metabolic control | 6 months
  To estimate the influence of the distribution of body mass and daily physical activity of patients with type 2 diabetes and SAHS on the metabolic response to treatment with CPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Garcia-Rio, MD, Study Chair — Hospital Universitario La Paz, IdiPAZ; Elizabet Martínez-Cerón, MD, Principal Investigator — Hospital Universitario La Paz, IdiPAZ; Alberto Alonso-Fernández, MD, Principal Investigator — Hospital Son Espasses
Locations (1):
- Hospital Universitario La Paz- IdiPaz, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Martinez-Ceron E, Barquiel B, Bezos AM, Casitas R, Galera R, Garcia-Benito C, Hernanz A, Alonso-Fernandez A, Garcia-Rio F. Effect of Continuous Positive Airway Pressure on Glycemic Control in Patients with Obstructive Sleep Apnea and Type 2 Diabetes. A Randomized Clinical Trial. Am J Respir Crit Care Med. 2016 Aug 15;194(4):476-85. doi: 10.1164/rccm.201510-1942OC. PMID 26910598